CLINICAL TRIAL: NCT02204137
Title: Pilot Study of the Falls Risk Questionnaire in Older Adults With Cancer
Brief Title: Falls Risk Questionnaire in Older Adults With Cancer
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201407080
Record Dates: First submitted 2014-07-23; First posted 2014-07-30 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Cancer; Geriatric Assessment
MeSH Terms: conditions — Neoplasms | interventions — ST13 protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Completion of Questionnaires: Participants will complete an assessment consisting of the Falls Risk Questionnaire, a primarily self-administered geriatric assessment (GA) developed by the Cancer and Aging Research Group, a quality of life scale (FACT GOG/NTX) and the Falls Efficacy Scale-International.
  Each questionnaire contains approximately 150 questions and will take between 30 minutes and one hour to complete.
  Interventions: Other: Falls Risk Questionnaire; Other: Cancer and Aging Research Group Geriatric Assessment; Other: Falls Efficacy Scale-International (FES-1); Other: Health Related Quality of Life using the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group Neurotoxicity Scale (FACT GOG/NTX)

INTERVENTIONS:
Other: Falls Risk Questionnaire
Other: Cancer and Aging Research Group Geriatric Assessment
Other: Falls Efficacy Scale-International (FES-1)
Other: Health Related Quality of Life using the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group Neurotoxicity Scale (FACT GOG/NTX)

SUMMARY:
The purpose of this research study is to look at the use of a series of questionnaires evaluating risk for falls in order to collect information that might be used to develop a larger study aiming to recognize who is more at risk for falls and how to best intervene to prevent falls in older adults with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older; 5 patients will be enrolled in each of the following age cohorts: 65-69, 70-74, 75-79, 80 and older
* Diagnosis of cancer, any type
* Currently receiving or anticipated to initiate systemic cancer therapy within 1 month, including endocrine therapy, chemotherapy or targeted therapies
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Unable to understand written English
* Psychiatric illness/social situation that would limit compliance with the study requirements
* Unable to walk.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cancer patients aged 65 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percent completion of the Fall Risk Questionnaire (FRQ) and the Cancer and Aging Research Group Geriatric Assessment (CARG GA) of enrolled patients | Day 1
  The percent of patients who complete the assessment will be calculated. Successful completion will be defined as the completion of all items on the questionnaires. If more than 85% of subjects are able to complete the FRQ and CARG GA, the assessment will be deemed feasible.

SECONDARY OUTCOMES:
Time to completion of FRQ and CARG GA of enrolled patients | Day 1
Satisfaction with the questionnaires | Day 1
  We will calculate the frequency of participant feedback that 1) certain questions that were difficult to understand 2) the questionnaire was too short or too long 3) questions were upsetting or 4) the questionnaire left out important questions to ask. Open-ended follow-up questions in which the participants will be given the opportunity to write out their responses will be examined qualitatively for recurring themes of particular questions that were unsatisfactory
Psychological consequences of falling | Day 1
  Uses the Falls Efficacy Scale-International (FES-I) and Health Related Quality of Life (HRQOL) using the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group Neurotoxicity Scale (FACT GOG/NTX)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Wildes, M.D., M.S.C.I., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu